CLINICAL TRIAL: NCT00787709
Title: Translational Research: Applying Drug Prevention to Obesity Prevention
Brief Title: Translational Obesity Research
Acronym: Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-08-00437; R01HD052107 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity prevention; Health promotion; School based curriculum
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Receives Pathways universal school-based health promotion curriculum from 4th-6th grade
  Interventions: Behavioral: Pathways
- 2 (No Intervention): Control group of students who do not receive the intervention

INTERVENTIONS:
Behavioral: Pathways — 3-year, 30 lesson, School-based universal health promotion curriculum with parent component.
  Arms: 1

SUMMARY:
The proposed project takes an innovative approach to childhood obesity prevention, for which there currently no evidence-based programs, and for which results of current trials have produced mainly short-term or disappointing effects. The aim of this project is to adapt and revise parts of two nationally recognized programs for drug prevention for use with children in grades 4-6 with the express purpose of obesity prevention. The current study will attempt to promote emotion regulation, neuro-cognitive function, and social competence in order to prevent obesity. A total of 24 elementary schools from two of the largest districts in Orange County will be randomly assigned to either the obesity prevention program or control group (N=1587) 4th grade students and their parents). A cohort of students will be followed from the 4th through 6th grades. Intervention students will be administered the Pathways obesity prevention program by trained teachers. The population is ethnically diverse (36% white, 57% Hispanic, 6%Asian; 48% on free/reduced lunch programs). Self-report measures, BMI, and waist circumference will be administered at the beginning of 4th grade, and at end of 4th , 5th , and 6th grade. Teacher, administrative, and parent surveys will be administered on the same schedule to measure school environment. Program implementation will be measured by teacher self-report and research staff observations. Data will be analyzed with statistical approaches that capture effects of school and classroom, test the theoretical model of change, and evaluate developmental trends in mediators and outcomes across the three grades. Findings should be generalizable to most elementary schools, and will be used to develop evidence-based program standards for childhood obesity prevention.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade students at participating schools

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Food Intake | 9 month posttest, 21 month follow-up, 33 month follow-up
Physical Activity | baseline, 9 month posttest, 21 month posttest, 33 month posttest
Body Mass Index | baseline, 9 month posttest, 21 month posttest, 33 month posttest

SECONDARY OUTCOMES:
Executive Cognitive Function | baseline, 9 month posttest, 21 month posttest, 33 month posttest
Stress | baseline, 9 month posttest, 21 month posttest, 33 month posttest
Attitudes toward healthy eating and physical activity | baseline, 9 month posttest, 21 month posttest, 33 month posttest

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Pentz, PhD, Principal Investigator — University of Southern California; Nathaniel R Riggs, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Alhambra, California, United States

REFERENCES:
- [Derived] Cappelli C, Pike JR, Christodoulou G, Riggs NR, Warren CM, Pentz MA. The effect of sensation seeking on alcohol use among middle school students: a latent state-trait analysis. Am J Drug Alcohol Abuse. 2020 May 3;46(3):316-324. doi: 10.1080/00952990.2019.1660885. Epub 2019 Sep 11. PMID 31509018
- [Derived] Cappelli C, Pike JR, Riggs NR, Warren CM, Pentz MA. Executive function and probabilities of engaging in long-term sedentary and high calorie/low nutrition eating behaviors in early adolescence. Soc Sci Med. 2019 Sep;237:112483. doi: 10.1016/j.socscimed.2019.112483. Epub 2019 Aug 7. PMID 31404882
- [Derived] Warren C, Riggs N, Pentz MA. Executive function mediates prospective relationships between sleep duration and sedentary behavior in children. Prev Med. 2016 Oct;91:82-88. doi: 10.1016/j.ypmed.2016.07.024. Epub 2016 Jul 29. PMID 27477059
- [Derived] Little MA, Riggs NR, Shin HS, Tate EB, Pentz MA. The effects of teacher fidelity of implementation of pathways to health on student outcomes. Eval Health Prof. 2015 Mar;38(1):21-41. doi: 10.1177/0163278713489879. Epub 2013 Jun 4. PMID 23739725
- [Derived] Pentz MA, Riggs NR. Longitudinal relationships of executive cognitive function and parent influence to child substance use and physical activity. Prev Sci. 2013 Jun;14(3):229-37. doi: 10.1007/s11121-012-0312-3. PMID 23345012
- [Derived] Pentz MA, Spruijt-Metz D, Chou CP, Riggs NR. High calorie, low nutrient food/beverage intake and video gaming in children as potential signals for addictive behavior. Int J Environ Res Public Health. 2011 Dec;8(12):4406-24. doi: 10.3390/ijerph8124406. Epub 2011 Nov 29. PMID 22408581